CLINICAL TRIAL: NCT02955927
Title: Combined Atropine With Orthokeratology in Childhood Myopia Control (AOK) -A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Pauline Cho, Prof, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20160406005/UW 16-404
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Myopia
Keywords: Myopia control,ortho-k, atropine eye drops, children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ortho-k and 0.01% atropine eye drops (Experimental): participants will receive treatment of ortho-k and 0.01% atropine eye drops
  Interventions: Drug: 0.01% atropine eye drops; Device: ortho-k
- ortho-k (Active Comparator): participants will receive treatment of ortho-k alone
  Interventions: Device: ortho-k

INTERVENTIONS:
Drug: 0.01% atropine eye drops
  Arms: ortho-k and 0.01% atropine eye drops
Device: ortho-k

SUMMARY:
This study aims to compare effects in retardation of myopia progression of combined ortho-k and 0.01% atropine therapy with those of ortho-k alone.Myopia control methods mainly focus on optical and pharmaceutical interventions . Currently, overnight-wear orthokeratology (ortho-k), is used extensively in Hong Kong with approximately 50% retardation effect. Pharmaceutical methods have focused on the use of atropine eye drops to slow myopic progression.The use of 1% atropine was limited by the manifestation of side effects and rebound effect.However, both side effect and rebound effect was minimal with 0.01% atropine.It was suggested that 0.01% was the optimum concentration for controlling myopia.The mechanisms of neither ortho-k nor atropine in myopia control are fully understood.It is believed that ortho-k and atropine act via different mechanisms.It is possible that by combining these two methods, additional retardation of myopia progression could be achieved.

DETAILED DESCRIPTION:
Although it is believed that myopia is the result of an interplay between genetic and environmental factors and its progression has been attributed to the lack of outdoor activities and intensive school work, myopia control methods mainly focus on optical and pharmaceutical interventions. Use of bifocal and multifocal lenses have been shown to be ineffective in myopia control. Specially designed soft contact lenses for myopia control have recently been launched, but their effectiveness has yet to be confirmed. Currently, overnight-wear orthokeratology (ortho-k), which involves reshaping the cornea by overnight wear allowing for improved, frequently unaided, vision during the day, is used extensively in Hong Kong. Approximately 50% retardation in axial length elongation was observed in studies of patients receiving ortho-k (LORIC study, 46%, ROMIO study,43%, and TO-SEE study, 52%).

Pharmaceutical methods have focused on the use of atropine eye drops to slow myopic progression. The use of 1% atropine was first suggested in the 1990's, but its application was limited by the manifestation of side effects such as pupil dilatation and loss of accommodation. The effectiveness of lower concentrations (0.5%, 0.1% and 0.01%) have been evaluated in a recent five-year randomized clinical trial, where the authors reported that 0.01% atropine once daily was effective resulting in about 50% of spherical equivalent reduction. However, this was as a result of one year (3rd year) discontinuation of atropine in the five-year study. Rebound effect was minimal with 0.01% atropine and higher dosages were associated with more manifest rebound effects, which appeared to negate former myopia retardation effects. Only 24% of those receiving 0.01% progressed 0.50D or more after discontinuation for one year. By contrast, proportion of children progressed 0.50D or more in 0.5% and 0.1% groups were 59% and 68% respectively. Moreover, use of 0.01% atropine showed sustained myopia reduction with clinically negligible effects on pupil dilatation and loss of accommodation. The authors suggested the use of 0.01% as the optimum concentration for controlling myopia.

The mechanisms of neither ortho-k nor atropine in myopia control are fully understood. It is believed that ortho-k and atropine act via different mechanisms, with ortho-k slowing myopia progression by reducing peripheral hyperopic defocus, while atropine exerts effects on anti-muscarinic receptors of the retina and sclera. However, some subjects respond poorly to either atropine or ortho-k, as demonstrated in clinical trials, suggesting that a single treatment may be not enough. It is possible that by combining these two methods, additional retardation of myopia progression could be achieved. In this randomized trial, we will explore the effectiveness of combination of ortho-k and atropine therapy, and evaluate additional effects by comparing the combination with ortho-k treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Manifest myopia between 1.00-4.00D in both eyes at screening visit
* Manifest astigmatism ≤2.50D; with-the-rule astigmatism (axes 180 ± 30) ≤2.50D; astigmatism with other axes ≤0.50D in both eyes at screening visit
* <1.00D difference in manifest spherical equivalent (SE) between the two eyes at screening visit
* Baseline cycloplegic objective refraction between 1.00-4.00D in sphere; astigmatism ≤2.50D; <1.00D difference in manifest SE between the two eyes
* Best-corrected logMAR visual acuity 0.10 or better in both eyes
* Symmetrical corneal topography with corneal toricity <2.00D in either eye
* Normal ocular health other than myopia
* Agree to be randomized and to attend the scheduled visits and aftercare

Exclusion Criteria:

* Contraindications to atropine: known allergies or cardiovascular disease, epilepsy
* Contraindications to contact lens wear and ortho-k: corneal scar, history of ocular inflammation/infection, limbus-to-limbus corneal cylinder and dislocated corneal apex
* Strabismus or amblyopia
* History of myopia control treatment (e.g. soft contact lenses, progressive add spectacles, atropine eye drops)
* Rigid contact lens (including ortho-k) wear experience
* Systemic condition which might affect refractive development (for example, Down syndrome, Marfan's syndrome)
* Ocular conditions which might affect refractive error (for example, cataract, ptosis)
* Poor response to lens wear including poor lens handling, poor vision and/ocular response after lens modifications
* Poor compliance with schedule visits

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Changes in axial length in 2 years | Every 6 months for a period of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Pauline, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Kowloon, Hong Kong

REFERENCES:
- [Background] Pan CW, Ramamurthy D, Saw SM. Worldwide prevalence and risk factors for myopia. Ophthalmic Physiol Opt. 2012 Jan;32(1):3-16. doi: 10.1111/j.1475-1313.2011.00884.x. PMID 22150586
- [Background] Lam CS, Lam CH, Cheng SC, Chan LY. Prevalence of myopia among Hong Kong Chinese schoolchildren: changes over two decades. Ophthalmic Physiol Opt. 2012 Jan;32(1):17-24. doi: 10.1111/j.1475-1313.2011.00886.x. PMID 22150587
- [Background] Fan DS, Lai C, Lau HH, Cheung EY, Lam DS. Change in vision disorders among Hong Kong preschoolers in 10 years. Clin Exp Ophthalmol. 2011 Jul;39(5):398-403. doi: 10.1111/j.1442-9071.2010.02470.x. Epub 2011 Feb 1. PMID 21105971
- [Background] Morgan IG, Ohno-Matsui K, Saw SM. Myopia. Lancet. 2012 May 5;379(9827):1739-48. doi: 10.1016/S0140-6736(12)60272-4. PMID 22559900
- [Background] Berntsen DA, Sinnott LT, Mutti DO, Zadnik K. A randomized trial using progressive addition lenses to evaluate theories of myopia progression in children with a high lag of accommodation. Invest Ophthalmol Vis Sci. 2012 Feb 13;53(2):640-9. doi: 10.1167/iovs.11-7769. Print 2012 Feb. PMID 22205604
- [Background] Correction of Myopia Evaluation Trial 2 Study Group for the Pediatric Eye Disease Investigator Group. Progressive-addition lenses versus single-vision lenses for slowing progression of myopia in children with high accommodative lag and near esophoria. Invest Ophthalmol Vis Sci. 2011 Apr 25;52(5):2749-57. doi: 10.1167/iovs.10-6631. PMID 21282579
- [Background] Paune J, Morales H, Armengol J, Quevedo L, Faria-Ribeiro M, Gonzalez-Meijome JM. Myopia Control with a Novel Peripheral Gradient Soft Lens and Orthokeratology: A 2-Year Clinical Trial. Biomed Res Int. 2015;2015:507572. doi: 10.1155/2015/507572. Epub 2015 Oct 28. PMID 26605331
- [Background] Cho P, Cheung SW, Edwards M. The longitudinal orthokeratology research in children (LORIC) in Hong Kong: a pilot study on refractive changes and myopic control. Curr Eye Res. 2005 Jan;30(1):71-80. doi: 10.1080/02713680590907256. PMID 15875367
- [Background] Cho P, Cheung SW. Retardation of myopia in Orthokeratology (ROMIO) study: a 2-year randomized clinical trial. Invest Ophthalmol Vis Sci. 2012 Oct 11;53(11):7077-85. doi: 10.1167/iovs.12-10565. PMID 22969068
- [Background] Chen C, Cheung SW, Cho P. Myopia control using toric orthokeratology (TO-SEE study). Invest Ophthalmol Vis Sci. 2013 Oct 3;54(10):6510-7. doi: 10.1167/iovs.13-12527. PMID 24003088
- [Background] Chua WH, Balakrishnan V, Chan YH, Tong L, Ling Y, Quah BL, Tan D. Atropine for the treatment of childhood myopia. Ophthalmology. 2006 Dec;113(12):2285-91. doi: 10.1016/j.ophtha.2006.05.062. Epub 2006 Sep 25. PMID 16996612
- [Background] Chia A, Chua WH, Cheung YB, Wong WL, Lingham A, Fong A, Tan D. Atropine for the treatment of childhood myopia: safety and efficacy of 0.5%, 0.1%, and 0.01% doses (Atropine for the Treatment of Myopia 2). Ophthalmology. 2012 Feb;119(2):347-54. doi: 10.1016/j.ophtha.2011.07.031. Epub 2011 Oct 2. PMID 21963266
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Brodstein RS, Brodstein DE, Olson RJ, Hunt SC, Williams RR. The treatment of myopia with atropine and bifocals. A long-term prospective study. Ophthalmology. 1984 Nov;91(11):1373-9. doi: 10.1016/s0161-6420(84)34138-0. PMID 6514306
- [Background] Liu Y, Wildsoet C. The effective add inherent in 2-zone negative lenses inhibits eye growth in myopic young chicks. Invest Ophthalmol Vis Sci. 2012 Jul 31;53(8):5085-93. doi: 10.1167/iovs.12-9628. PMID 22761258
- [Background] Arumugam B, McBrien NA. Muscarinic antagonist control of myopia: evidence for M4 and M1 receptor-based pathways in the inhibition of experimentally-induced axial myopia in the tree shrew. Invest Ophthalmol Vis Sci. 2012 Aug 24;53(9):5827-37. doi: 10.1167/iovs.12-9943. PMID 22836762
- [Derived] Tan Q, Ng AL, Choy BN, Cheng GP, Woo VC, Cho P. One-year results of 0.01% atropine with orthokeratology (AOK) study: a randomised clinical trial. Ophthalmic Physiol Opt. 2020 Sep;40(5):557-566. doi: 10.1111/opo.12722. Epub 2020 Aug 10. PMID 32776533